## Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

Protocol Title: Clinical Evaluation of etafilcon A Contact Lenses Using a Novel

Manufacturing Technology

Protocol CR-6324

Version: 2.0, Amendment 1.0

Date: April 26, 2019

Investigational Products: etafilcon A

Key Words: Words: etafilcon A, mold process, daily disposable

## Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

## TABLE OF CONTENTS

| SPONS | SOR NAME AND ADDRESS | 6 |
|---|---|---|
| MEDIC | CAL MONITOR | 6 |
| AUTHO | ORIZED SIGNATURES | 7 |
| CHANG | GE HISTORY | 8 |
| SYNOI | PSIS | 9 |
| COMM | MONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 1. IN | TRODUCTION AND BACKGROUND | 16 |
| 1.1. | Name and Descriptions of Investigational Products | 16 |
| 1.2. | Intended Use of Investigational Products | 16 |
| 1.3. | Summary of Findings from Nonclinical Studies | 16 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 16 |
| 1.5.<br>Clini | Relevant Literature References and Prior Clinical Data Relevant to ical Study | - |
| 2. ST | TUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 16 |
| 2.1. | Objectives | 16 |
| 2.2. | Endpoints | 17 |
| 2.3. | Hypotheses | 18 |
| 3. TA | ARGETED STUDY POPULATION | 18 |
| 3.1. | General Characteristics | 18 |
| 3.2. | Inclusion Criteria | 19 |
| 3.3. | Exclusion Criteria | 19 |
| 3.4. | Enrollment Strategy | 20 |
| 4. ST | TUDY DESIGN AND RATIONALE | 20 |
| 4.1. | Description of Study Design | 20 |
| 4.2. | Study Design Rationale | 21 |
| 4.3. | Enrollment Target and Study Duration | 21 |
| 5. TE | EST ARTICLE ALLOCATION AND MASKING | 22 |
| 5.1. | Test Article Allocation | 22 |
| 5.2. | Masking | 22 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 23 |
| 6. ST | TUDY INTERVENTION | 23 |
| 6.1. | Identity of Test Articles | 23 |
| 6.2. | Ancillary Supplies/Products | 24 |

| 6. | 3. | Administration of Test Articles | 24 |
|---|---|---|---|
| 6. | 4. | Packaging and Labeling | 24 |
| 6 | 5. | Storage Conditions | 25 |
| 6. | 6. | Collection and Storage of Samples | 25 |
| 6. | 7. | Accountability of Test Articles | 25 |
| 7. | STU | JDY EVALUATIONS | 26 |
| 7. | 1. | Time and Event Schedule | 26 |
| 7. | 2. | Detailed Study Procedures | 27 |
| | VIS | IT 1 | 27 |
| | VIS | IT 2 | 32 |
| | VIS | IT 3 | 34 |
| | VIS | IT 4 | 38 |
| | FIN | AL EVALUATION | 40 |
| 7. | | Unscheduled Visits | |
| 7. | 4. | Laboratory Procedures | 41 |
| 8. | SUI | BJECTS COMPLETION/WITHDRAWAL | 41 |
| 8. | 1. | Completion Criteria | 41 |
| 8. | 2. | Withdrawal/Discontinuation from the Study | 41 |
| 9. | PRI | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 42 |
| 10. | D | EVIATIONS FROM THE PROTOCOL | 42 |
| 11. | S | ΓUDY TERMINATION | 43 |
| 12. | Pl | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 43 |
| 13. | A | DVERSE EVENTS | 45 |
| 13 | 3.1. | Definitions and Classifications | 45 |
| 13 | 3.2. | Assessing Adverse Events | 47 |
| | 13.2 | 2.1. Causality Assessment | 47 |
| | 13.2 | 2.2. Severity Assessment | 48 |
| 13 | 3.3. | Documentation and Follow-Up of Adverse Events | 48 |
| 13 | 3.4. | Reporting Adverse Events | 49 |
| | 13.4 | 4.1. Reporting Adverse Events to Sponsor | 49 |
| | 13.4<br>Aut | 4.2. Reporting Adverse Events to the Responsible IEC/IRB and Industries | |
| | 13.4 | 4.3. Event of Special Interest | 50 |
| 13 | 3.5. | Reporting of Pregnancy | 50 |
| 1/1 | Q" | TATISTICAL METHODS | 51 |

| 14. | .1. | General Considerations. | 51 |
|---|---|---|---|
| 14. | .2. | Sample Size Justification | 51 |
| 14. | .3. | Analysis Populations | 52 |
| 14. | .4. | Level of Statistical Significance | 53 |
| 14. | .5. | Primary Analysis | 53 |
| 14. | .6. | Secondary Analysis | 53 |
| 14. | .7. | Other Exploratory Analyses | 54 |
| 14. | .8. | Interim Analysis | 54 |
| 14. | .9. | Procedure for Handling Missing Data and Drop-Outs | 54 |
| 14. | .10. | Procedure for Reporting Deviations from Statistical Plan | 55 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 55 |
| 15. | .1. | Electronic Case Report Form/Data Collection | 55 |
| 15. | .2. | Subject Record | 55 |
| 16. | DA | TA MANAGEMENT | 56 |
| 16. | .1. | Access to Source Data/Document | 56 |
| 16. | .2. | Confidentiality of Information. | 56 |
| 16. | .3. | Data Quality Assurance | 56 |
| 17. | MO | NITORING | 57 |
| 18. | ETI | HICAL AND REGULATORY ASPECTS | 57 |
| 18. | .1. | Study-Specific Design Considerations | 57 |
| 18. | .2. | Investigator Responsibility | 57 |
| 18. | .3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 58 |
| 18. | .4. | Informed Consent | 59 |
| 18. | .5. | Privacy of Personal Data | 60 |
| 19. | STU | JDY RECORD RETENTION | 61 |
| 20. | FIN | ANCIAL CONSIDERATIONS | 61 |
| 21. | PUl | BLICATION | 62 |
| 22. | REI | FERENCES | 62 |
| | | X A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | |
| APPI | ENDI | X B: PATIENT INSTRUCTION GUIDE | 70 |
| APPI | ENDI | X C: PACKAGE INSERT (APPROVED PRODUCT) | |
| APPI | ENDI | X D: | |
| | | LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS | 101 |
| | | EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | 109 |

| LENS FITTING CHARACTERISTICS |
|---|
| SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS 121 |
| FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE 123 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS |
| BIOMICROSCOPY SCALE |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION 142 |
| DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE |
| PATIENT REPORTED OUTCOMES |
| WHITE LIGHT LENS SURFACE WETTABILITY |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE 161 |
| TABLE OF CONTENTS Figure 1: Study Flowchart |
| TABLE OF CONTENTS |
| Table 1: Target number of subjects by arm and phase |
| Table 3: Ancillary Supplies |
| Table 4: Time and Events |
| Table 5: 1-week CLUE comfort and vision for 1 Day ACUVUE MOIST in historical studies |
| Table 6: Power Analysis for CLUE scores |

## PROTOCOL TITLE, NUMBER, VERSION

Title: Clinical Evaluation of etafilcon A Contact Lenses Using a Novel Manufacturing

Technology

Protocol Number: CR-6324 Version: 2.0, Amendment 1.0

Date: April 26, 2019

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR

Name: Brian Pall, OD, MS, FAAO

Title: Senior Principal Research Optometrist

Address: 7500 Centurion Parkway, Suite 100, Mail W-2A, Jacksonville, FL 32256

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| See Electronic Signature Report Brian Pall, OD, MS, FAAO Sr. Principal Research Optometrist | DATE |
|---|---|
| See Electronic Signature Report | DATE |
| See Electronic Signature Report | DATE |
| See Electronic Signature Report | DATE |
| See Electronic Signature Report | DATE |
| See Electronic Signature Report | DATE |
| | Brian Pall, OD, MS, FAAO Sr. Principal Research Optometrist See Electronic Signature Report See Electronic Signature Report See Electronic Signature Report See Electronic Signature Report |

## **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | Brian Pall | Original Protocol | December 20, 2018 |
| 2.0 | Brian Pall | <ul> <li>Section 4.1: Remove "group sequential" from the study design description</li> <li>Section 14.2: Change "5% confidence level" to "5% significance level"</li> <li>General protocol clarifications <ul> <li>Temperature monitoring of refrigerator not required</li> <li>Multiple brands of sterile rewetting drops listed</li> <li>Protocol duration will be approximately 7 weeks</li> <li>Patient visits that are out of window at Visits 2 and 4 will be excluded from the cohort population</li> </ul> </li> </ul> | April 26, 2019 |

## **SYNOPSIS**

| Protocol Title | Clinical Evaluation of etafilcon A Contact Lenses Using a |
|---|---|
| | Novel Manufacturing Technology |
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Phase 0: Feasibility Study |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the |
| | Sponsor |
| Test Article(s) | <b>Investigational Products:</b> |
| | • etafilcon A contact lenses made with a novel |
| | manufacturing technology (Test) |
| | • etafilcon A contact lenses made with the current |
| | manufacturing technology (Control). |
| Wear and Replacement | Wear Schedule: daily wear |
| Schedules | Replacement Schedule: daily disposable |
| Objectives | To evaluate the clinical performance of etafilcon A contact |
| | lenses made with a new manufacturing technology as |
| | compared to etafilcon A contact lenses made with the existing |
| | manufacturing technology. |
| Study Endpoints | Co-primary endpoint(s): |
| | <ul> <li>Overall comfort after 1-week of lens wear</li> </ul> |
| | <ul> <li>Overall quality of vision after 1-week of lens wear</li> </ul> |
| | Secondary endpoint(s): |
| | <ul> <li>Monocular distance visual performance</li> </ul> |
| | <ul> <li>Average daily wear time (in hour)</li> </ul> |
| | Additional Endpoints: |
| | Slit lamp findings |
| | <ul> <li>Subject reported ocular symptoms</li> </ul> |
| | <ul> <li>Lens fitting characteristics</li> </ul> |
| | Lens wettability |
| | Adverse events |
| Study Design | This study is a feasibility, multi-site, randomized, double- |
| | masked, 2×2 crossover design, 1-week dispensing study. |
| | Subjects will wear bilaterally both Test and Control lenses in a |
| | random order for 1-week each as a daily disposable modality |
| | with a wash-out period of 1 week between the wearing |
| | periods. |
| | See the flow chart at the end of the synopsis table for the |
| | schematic of the study visits and procedures of main |
| G 1 G' | observations (Figure 1). |
| Sample Size | Up to 100 eligible subjects will be enrolled and randomized |
| | into the study to ensure that approximately 90 subjects |
| | complete as cohort. |

| Study Duration | The study will last approximately 7 weeks and include an enrollment period of 3 weeks. |
|---|---|
| Anticipated Study<br>Population | Healthy male and female volunteers (at least 18 and not more than 70 years old) who are habitual wearers of daily disposable contact lenses (approximately 80% 1-Day ACUVUE Moist, approximately 20% other daily disposable hydrogel contact lens brands) and have a spectacle astigmatism of <0.75D in both eyes. |
| Eligibility Criteria | Potential subjects must satisfy all of the following criteria to be enrolled in the study: Inclusion Criteria after Screening |
| | <ol> <li>The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Must be at least 18 and not more than 70 years of age (including 70) at the time of screening.</li> <li>The subject must be a habitual and adapted wearer of hydrogel daily disposable brand contact lenses in both eyes (at least 1 month of daily wear).</li> <li>The subject must have normal eyes (i.e., no ocular medications or infections of any type).</li> </ol> |
| | <ul> <li>6. The subject's required spherical contact lens prescription must be in the range of -0.50 to -6.00 D in each eye.</li> <li>7. The subject's refractive cylinder must be &lt; 0.75D in each eye.</li> <li>8. The subject must have best corrected visual acuity of 20/25 or better in each eye.</li> </ul> |
| | Exclusion Criteria after Screening |
| | Potential subjects who meet any of the following criteria will be excluded from participating in the study: 1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued). 2. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear. 3. Any previous, or planned, ocular or interocular surgery |

| | (e.g., radial keratotomy, PRK, LASIK, etc.). |
|---|---|
| | 4. Any ocular infection. |
| | 5. Any corneal distortion resulting from previous hard or |
| | rigid gas permeable contact lens wear. |
| | 6. Monovision or multi-focal contact lens correction. |
| | 7. Participation in any contact lens or lens care product |
| | clinical trial within 14 days prior to study enrollment. 8. History of binocular vision abnormality or strabismus. |
| | 9. Any infectious disease (e.g., hepatitis, tuberculosis) or |
| | a contagious immunosuppressive disease (e.g., HIV, by |
| | self-report). |
| | 10. Suspicion of or recent history of alcohol or substance |
| | abuse. |
| | 11. History of serious mental illness. |
| | 12. History of seizures. |
| | 13. Employee or immediate family member of an |
| | employee of clinical site (e.g., Investigator, |
| | Coordinator, Technician) |
| | Exclusion Criteria after Baseline |
| | 14. Any ocular allergies, infections or other ocular |
| | abnormalities that are known to interfere with contact |
| | lens wear and/or participation in the study. This may |
| | include, but not be limited to entropion, ectropion, |
| | extrusions, chalazia, recurrent styes, glaucoma, history |
| | of recurrent corneal erosions, aphakia, or corneal |
| | distortion |
| | 15. Any Grade 3 or greater slit lamp findings (e.g., edema, |
| | corneal neovascularization, corneal staining, tarsal |
| | abnormalities, conjunctival injection) on the Food and |
| | Drug Administration (FDA) classification scale |
| | 16. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer |
| | or round peripheral scar), or any other ocular |
| | abnormality that may contraindicate contact lens wear. |
| Disallowed | Disallowed medications include any medication that may |
| Medications/Interventions | interfere with contact lens wear (at the investigator's |
| | discretion). |
| Measurements and | Subjective assessments, physiological responses, fitting |
| Procedures | characteristics. |
| Microbiology or Other | None |
| Laboratory Testing | |

| Study Termination | The occurrence of one or more Unanticipated Adverse Device |
|---|---|
| | Effect (UADE), or any SAE where relationship to study agent |
| | cannot be ruled out, will result in stopping further dispensing |
| | investigational product. In the event of a UADE or SAE, the |
| | Sponsor Medical Monitor may unmask the treatment regimen |
| | of subject(s) and may discuss this with the Principal |
| | Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | Sterile rewetting drops |
| Specific Materials | |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Study Flowchart

Biomicroscopy
Patient Instructions



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience
COM Clinical Operations Manager
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CWT Comfortable Wear Time

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HLLC High Luminance With Low Contrast Charts

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IEC Independent Ethics Committee IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LASIK Laser-Assisted In Situ Keratomileusis

LLHC Low Luminance With High Contrast Charts

LogMAR Logarithm of Minimal Angle of Resolution MPMVA Maximum Plus To Maximum Visual Acuity

OD Right Eye
OS Left Eye
OU Both Eyes

PD Protocol Deviation
PI Principal Investigator
PIG Patient Instruction Guide
PP Predictive Probability
PQC Product Quality Complaint
PRK Photorefractive Keratectomy
PRO Patient Reported Outcome

QA Quality Assurance

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity WT Wear Time

#### 1. INTRODUCTION AND BACKGROUND

In the spirit of continuous improvement, JJVC has identified a new manufacturing technology for etafilcon A. The purpose of this clinical trial is to demonstrate whether this new manufacturing technology has any clinically relevant impact on the clinical performance of the contact lens.

## 1.1. Name and Descriptions of Investigational Products

The investigational products are:

- etafilcon A contact lenses made with a new manufacturing technology (Test).
- etafilcon A contact lenses made with the current manufacturing technology (Control).

## 1.2. Intended Use of Investigational Products

The intended use of the investigative products is for correcting refractive error. During the study, each test article will be worn bilaterally in daily wear, daily disposable modality for at least 8 hours per day for approximately 1 week.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding etafilcon A refer to the latest version of the Investigator's Brochure (IB).

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

For the most comprehensive risk and benefit information regarding etafilcon A product refer to the latest version of the Investigator's Brochure (IB).

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

See Package Inserts for 1-DAY ACUVUE® MOIST. (APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT).

## 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

Primary Objective(s)

To evaluate the clinical performance of etafilcon A contact lenses made with a new manufacturing technology as compared to etafilcon A contact lenses made with the existing manufacturing technology in the following areas:

- Overall comfort.
- Overall quality of vision

#### Secondary Objective(s)

To evaluate the clinical performance of etafilcon A lenses made with a new manufacturing technology by comparison to etafilcon A lenses made with the manufacturing technology in the following areas:

- Monocular distance visual performance (in logMAR)
- Average daily wear time (in hours)

## 2.2. Endpoints

## **Primary Endpoint(s)**

#### CLUE Comfort and Vision Scores:

The co-primary endpoints for this study are subjective assessment of comfort and quality of vision after 7±2 days of wearing the study lenses as a daily disposable.

Subjective assessment of comfort and vision will be performed using the Contact Lens User Experience<sup>TM</sup> (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire used to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a US contact-lens wearing population between 18 and 65 years of age. CLUE composite scores are derived using Item Response Theory (IRT) and follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for the population of soft disposable contact lens wearers.

## Secondary Endpoint(s)

## Average daily wear time (in hours):

Average daily wear time will be calculated as the number of hours between subjects reported time of insertion and time of removal of the study lenses, on an average day, at 1-Week Follow up evaluation.

#### Visual performance

Visual performance will be calculated as monocular contact lens-corrected distance visual acuity using a logMAR visual acuity scale. This will be evaluated under both high luminance/low contrast conditions and low luminance/high contrast conditions at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts at the 1 Week Follow-up visit.

#### Other Endpoint(s)

## Slit Lamp Findings

Frequency and severity by eye of slit lamp findings (SLFs) including conjunctival injection, corneal edema, corneal neovascularization, corneal staining, tarsal abnormalities or any other complications. SLFs will be evaluated at fitting and post-fitting evaluation visits including unscheduled visits.

## Subject's Reported Ocular Symptoms

Frequency and severity by eye of subject's reported ocular symptoms and problems with the study lens at fitting and post-fitting evaluation visits including unscheduled visits.

#### Lens Fitting characteristics

Frequency by eye of mechanical lens fitting characteristics including lens centration and lens movement and overall lens fitting acceptability at fitting and 1-week follow-up evaluations.

#### Lens wettability:

Frequency and Grade by eye of lens wettability at 1-Week Follow-up evaluation.

The following will be monitored and descriptively evaluated

- Adverse events
- Reasons for discontinuation
- Lens damage

#### 2.3. Hypotheses

This is a feasibility study and all the hypotheses are exploratory in nature.

## Primary Hypotheses:

There are two co-primary hypotheses in this study. Both of them must be met to satisfy the primary objective of the study.

- 1. The Test lens will be non-inferior to the Control lens with respect to overall CLUE comfort score at the follow-up visit. A non-inferiority margin of -5 points will be used.
- 2. The Test lens will be non-inferior to the Control lens with respect to overall CLUE vision score at the follow-up visit. A non-inferiority margin of -5 points will be used.

## **Secondary Hypotheses:**

- 1. The Test lens will be non-inferior to the Control lens with respect to logMAR visual performance (using ETDRS visual acuity charts) at the follow-up visit. A non-inferiority margin of 0.05 logMAR will be used.
- 2. The Test lens will be non-inferior to the Control lens with respect to average daily wear time at 1-week follow-up visit. A non-inferiority margin of 1 hour will be used.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

The population to be studied will be healthy male and female volunteers (at least 18 and not more than 70 years old) who are habitual wearers of daily disposable (approximately 80% 1 Day ACUVUE MOIST, approximately 20% any other brand of hydrogel daily disposable

contact lens) and have a spectacle astigmatism of <0.75 D in both eyes. Up to 100 subjects will be enrolled to ensure approximately 90 subjects successfully complete the study.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

## Inclusion Criteria after Screening

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Must be at least 18 and not more than 70 years of age (including 70) at the time of screening.
- 4. The subject must be a habitual and adapted wearer of hydrogel daily disposable brand contact lens in both eyes (at least 1 month of daily wear).
- 5. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

#### Inclusion Criteria after Baseline

- 6. The subject's required spherical contact lens prescription must be in the range of -0.50 to -6.00 D in each eye.
- 7. The subject's refractive cylinder must be < 0.75 D in each eye.
- 8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

#### Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
- 2. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
- 3. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 4. Any ocular infection.
- 5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
- 6. Monovision or multi-focal contact lens correction.
- 7. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
- 8. History of binocular vision abnormality or strabismus.

- 9. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self-report).
- 10. Suspicion of or recent history of alcohol or substance abuse.
- 11. History of serious mental illness.
- 12. History of seizures.
- 13. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician)

#### Exclusion Criteria after Baseline

- 14. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
- 15. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale.
- 16. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.

## 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

## 4.1. Description of Study Design

This study is a multi-site, randomized, double-masked,  $2\times2$  crossover design, 1-week dispensing study. Subjects will wear bilaterally both Test and Control lenses in a random order for 1-week each as a daily disposable modality with a wash-out period of 1 week between the wearing periods.

#### Period 1:

At study Visit 1, subjects\_will be consented and screened for inclusion/exclusion criteria. If a subject is found to meet all eligibility criteria (see Section 3.4.), they will be randomly assigned to either Test/Control or Control/Test sequence using 1:1 ratio (i.e. 1/2 of subjects on the Test/Control sequence and 1/2 on the Control/Test sequence). Subjects will fit the first pair of lens in both eyes based on the sequence assigned; otherwise, the subject will be deemed ineligible for this study. Subjects will be advised to wear the study lenses at least 8 hours a day for a minimum of 5 days.

Successfully dispensed subjects at the Visit 1 will be scheduled for a follow-up visit (Visit 2). The follow-up visit will occur approximately 7±2 days after the Visit 1. Unscheduled follow-up visits may occur during the study. At this visit, CLUE comfort and vision, slit lamp findings will be captured.

#### Wash-out period:

After completion of Visit 2, there is a 7 to 9 day washout period during which subjects may use their habitual products.

#### Period 2:

Following the washout period, the subject returns for Visit 3 and post-washout baseline evaluation will take place prior to lens fitting. After baseline evaluation, subject will be fitted and dispensed with the second pair of lens in the assigned sequence. Subjects will be advised to wear the study lenses at least 8 hours a day for a minimum of 5 days.

Visit 4 takes place 7±2 days after Visit 3, at which CLUE comfort and vision, slit lamp findings, final evaluation will take place.

Both study lenses will be worn as a daily disposable modality. JJVC will provide the investigational sites with sufficient quantities of study lenses and supplies to complete the study.

#### 4.2. Study Design Rationale

The crossover study design will allow each subject to evaluate both the Test and Control lenses and will help to reduce potential intra-subject variation. To reduce any potential carryover effect, a 7 to 9 day washout period was considered between the wearing periods.

Both lenses will be worn as daily disposable modality, therefore 1-week wearing period was considered sufficiently longer to assess the primary and secondary objectives of the study.

## 4.3. Enrollment Target and Study Duration

Up to 100 subjects will be initially enrolled and approximately 90 are targeted to complete the study.

The population to be studied will be healthy male and female volunteers (at least 18 and not more than 70 years old) who are habitual wearers of daily disposable (approximately 80% 1 Day ACUVUE MOIST, approximately 20% any other brand of hydrogel daily disposable contact lens) and have a spectacle astigmatism of <0.75 D in both eyes.

The Investigator is responsible for ensuring that all subjects entering the study conform to subject selection criteria. The number of subjects targeted for randomization and completion are as follows:

Table 1: Target number of subjects by arm and phase

| | Test/Control | Control/Test | Total |
|-------------------------|--------------|--------------|-------|
| Randomization | 50 | 50 | 100 |
| Completion | 45 | 45 | 90 |
| Number of sites | 6 | 6 | 6 |
| Subjects/site (Min-Max) | 5-10 | 5-10 | 10-20 |

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2×2 crossover design. A computer-generated randomization scheme will be used to randomly assign subjects, in block of 2, to one of the two possible lens wear sequences: Test/Control or Control/Lens. The random scheme will be generated using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment per the randomization list and not pre-select or assign subjects. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected.

#### 5.2. Masking

This is a double-masked study where subjects, investigators are masked to the identity of the study lenses during the study period. Every attempt will be made to keep the other clinical trial personnel involved in the study (e.g. data management, biostatistician) unaware of the identity of the study lenses.

The identity of the study lenses will be masked by over labeling the blister packs with a label containing the study number, lot number, sphere power, expiration date and the randomization codes. Only the personnel involved in the over labeling and the statistician generating the randomization scheme will have access to the decode information translating the randomization codes into Test and Control groups. The Biostatistician performing the interim analysis will have access to the decode information to run the interim analysis. The medical monitor will also have access to the decode information in case breaking the mask is necessary for the urgent medical treatment of a subject.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken

only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued will not be replaced.

## 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken. The Biostatistician performing the interim analysis should keep the decode information in a secure location and should not share it with the personnel involved in the study until the all subjects have completed the study and the database is finalized.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- Investigator or designee (documented on the Delegation Log) will consult the lens
  fitting schedule/randomization scheme to obtain the test article assignment for that
  subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 2: Test Articles

| | Test | Control |
|--------------|--------------------------|--------------------------|
| Name | etafilcon A with novel | etafilcon A with current |
| | manufacturing technology | manufacturing |
| | | technology |
| Manufacturer | JJVC – 5GT | JJVC – 4GT |
| | | 1993 |

| . [ | Test | Control |
|---|---|---|
| Len Material | etafilcon A | etafilcon A |
| Nominal Base Curve @ 22 °C | 8.5 | 8.5 |
| Nominal Diameter @ 22 °C | 14.2 | 14.2 |
| Nominal Distance Powers (D) | -0.50 to -6.00<br>in 0.25 steps | -0.50 to -6.00<br>in 0.25 steps |
| Wear Schedule in Current Study | Daily wear | Daily wear |
| Replacement Frequency | Daily disposable | Daily disposable |
| Packaging Form (vial, blister, etc.) | Sterile blister pack | Sterile blister pack |

## 6.2. Ancillary Supplies/Products

The Sponsor will provide sterile rewetting drops for subject use if needed to relieve dryness. Subjects should not use their habitual rewetting drops during the study.

The following solutions may be used in this study:

Table 3: Ancillary Supplies

| | Solution |
|---------------------------|-----------------------------------------------|
| Solution Name/Description | Single use EyeCept or LacriPure or ScleralFil |
| Manufacturer | OPTICS Laboratory Inc/Menicon/ B+L |
| Preservative | None |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

## 6.4. Packaging and Labeling

The test articles will be packaged in blisters as the primary packaging. The test article will be over-labeled to mask the subject/Investigators to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



#### **6.5.** Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

## 6.6. Collection and Storage of Samples

Lenses that are being collected will be stored wet (using saline solution) in separate glass vials with labels that minimally contain study number, date, subject number, and eye from which the lens was removed.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

## 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

## 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 4: Time and Events

| | | isit 1<br>Pay 0) | Visit 2<br>(Day 5-9<br>from Visit 1) | (After a | sit 3<br>7-9 day<br>at period) | Visit 4<br>(Day 5-9<br>from Visit 3) |
|---|---|---|---|---|---|---|
| Estimated Visit<br>Duration | 1.5 H | Iours | 1 Hour | 1 Hour | | 1 Hour |
| Event | Baseline | Trial #1<br>Dispense | Trial #1<br>Follow-up Visit | Post<br>Washout<br>Baseline | Trial #2<br>Dispense | Trial #2<br>Follow-up<br>Visit and Exit |
| Study Informed<br>Consent | X | | | | | |
| Demographics | X | | | | | |
| Medical History | X | | | X | | |
| Eligibility<br>Assessment | X | | | X | | |
| Background<br>Questionnaire | X | | i i | | | |
| Subject Reported<br>Symptoms | X | X | X | X | X | X |
| Distance Visual<br>Acuity | X | X | X | X | X | X |
| Spherocylindrical<br>Refraction & VA | X | | | | | |
| Biomicroscopy &<br>Eye Rinse | X | | X | X | | X |
| Study Lenses<br>Dispensed | | X | | | X | |
| Lens Damage | | X | X | | X | X |
| Spherical Over-<br>Refraction | | X | | | X | |
| logMAR visual<br>acuity (ETDRS<br>charts) | | X | X | | X | X |
| Lens Fit<br>Assessment | | X | X | | X | X |
| Lens Surface<br>Deposits & Lens<br>Wettability<br>Assessment | | X | X | | X | X |

| | | sit 1<br>ay 0) | Visit 2<br>(Day 5-9<br>from Visit 1) | (After a | it 3<br>7-9 day<br>t period) | Visit 4<br>(Day 5-9<br>from Visit 3) |
|---|---|---|---|---|---|---|
| Estimated Visit<br>Duration | 1.5 Hours | | 1 Hour | 1 Hour | | 1 Hour |
| Event | Baseline | Trial #1<br>Dispense | Trial #1<br>Follow-up Visit | Post<br>Washout<br>Baseline | Trial #2<br>Dispense | Trial #2<br>Follow-up<br>Visit and Exit |
| Compliance | | | X | | | X |
| Contact Lens Wear<br>Time | X | | X | X | | X |
| Follow-up<br>Questionnaire | | | X | | | X |
| Adverse Event<br>Review | | | X | | | X |
| Concomitant<br>Medication<br>Review | X | | X | X | | X |
| Study Completion | | | | | | X |

## 7.2. Detailed Study Procedures

## VISIT 1

Screening Visit, Baseline Evaluation, Dispensing Visit.

Subjects should attend wearing their habitual lenses.

| Suoje | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of Informed<br>Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's year of birth, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |

| | | Visit 1: Screening | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters | |
| 1.5 | Contact lens wear times | Record the current wear time (WT) and comfortable wear time (CWT). | |
| 1.6 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must<br>be answered "yes" and all responses to Exclusion<br>Criteria questions must be answered "no" for the<br>subject to be considered eligible.<br>If subject is deemed to be ineligible after<br>screening, proceed to Final Evaluation and<br>complete all forms. | |
| ~ | | Visit 1: Baseline | Table 1 |
| Step | Procedure | Details | |
| 1.7 | Background PRO<br>Questionnaire (CLUE) | Subject will complete questions regarding their experiences with their habitual lenses. | |
| 1.8 | Subject-reported<br>Ocular Symptoms | Subject Reported Ocular Symptoms and Problems | |
| 1.9 | Distance visual acuity (VA) | Record the distance Snellen VA for OD, OS and OU. Subject must keep reading smaller lines until less than half the letters are correctly identified. | |
| 1.10 | Remove habitual lenses | The subject's habitual lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. | |
| 1.11 | Subjective<br>spherocylinder<br>refraction and VA | Perform binocular subjective best spherocylinder refraction and record the best corrected VA for OD, OS and OU. | |
| 1.12 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are Grade 3 or higher, the subject is discontinued from the visit as ineligible and may be rescheduled for another baseline visit for the randomization period. | |
| | | Limbal and Bulbar Conjunctival Hyperemia findings and detailed Corneal Staining Assessment will be recorded using a more detailed scale for internal purposes only. Conjunctival hyperemia should be assessed using the 0.5 increment grading scale. | |
| 1.13 | Eye Rinse | The investigator or technician may rinse the subject's eyes thoroughly with sterile saline. | |

| | | Visit 1: Baseline | au- |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.14 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. One additional baseline examination is permitted to be performed if the subject does not meet the eligibility criteria at the initial baseline visit If subject is deemed to be ineligible after baseline, proceed to Final Evaluation and complete all forms. | |
| d- | | Visit 1: Treatment 1 | |
| Step | Procedure | Details | |
| 1.15 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective best sphere refraction. Record the test condition. | |
| 1.16 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Note: A Patient Instruction Guide (PIG) will be given to the subject in any study where a lens is placed on eye. The subject may wear the study lenses only at the clinical site, or the subjects may be dispensed additional lenses to wear outside of the clinical site. | |
| 1.17 | Lens Damage | Using the slit lamp, assess lenses for damage. If any defects are noted, investigator should complete a Product Quality Complaint in EDC. Damaged lenses will be removed and stored in the following manner: The OD and OS lenses will be stored wet (using saline solution) in separate glass vials with labels that minimally contain study number, date, subject number, and eye from which the lens was removed. Replace lens if damaged. | |
| 1.18 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 1.19 | Subjective Best Sphere<br>Over Refraction | Perform subjective best sphere refraction over the study lenses with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) | |

| | Visit 1: Treatment 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS, and OU). | |
| | | Note: The endpoint criterion for the duo-chrome test is the lens power at which the red and green sides of the chart appear to be equally distinct. However, if the subject's response changes from "red" to "green" with only a 0.25D change in power and no report that the two sides appear to be equally sharp, the refraction endpoint should be the lens power that leave the red chart sharper. | |
| 1.20 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is not plano. For each power modification, repeat steps (1.15-1.19). | |
| | C 1: . P 1 | Up to one power modifications is allowed. | |
| 1.21 | Subject Reported | Subjects will respond to a verbal open-ended | FD1 -203 |
| 1.22 | Ocular Symptoms Subjective Lens Fit Assessment | symptoms questionnaire. Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. | |
| | | An unacceptable fit is deemed by one of the following criteria: • limbal exposure at primary gaze or with extreme eye movement • edge lift | |
| | | <ul> <li>excessive movement in primary and up gaze</li> <li>insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up</li> <li>Note: if lens fit is unacceptable subject will be</li> </ul> | |
| | | discontinued from the study. | |
| 1.23 | Distance ETDRS LogMAR Visual Acuity | Perform monocular distance ETDRS LogMAR visual acuity test at a 4-meter distance over the test eye only under the following conditions: | |
| | | <ul> <li>dim illumination (e.g., &lt;2.5 lux), low luminance, with high contrast charts (LLHC)</li> <li>bright illumination (e.g., &gt;400 lux), high</li> </ul> | |

| | Visit 1: Treatment 1 | |
|---|---|---|
| Step | Procedure | Details |
| | 11000000 | luminance with low contrast charts (HLLC) |
| | | The Precision Vision 4-meter high contrast ETDRS charts (Chart 1 and Chart 2 OD, Chart 3 and Chart 4 OS) and low contrast ETDRS charts (Chart 1 and 2 OD and Chart 3 and Chart 4 OS) will be used. |
| | | Two measurements per condition will be performed. |
| 1.24 | White Light Lens<br>Surface Wettability | Record the white light lens wettability of both lenses. |
| 1.25 | Surface Deposits | Record any front and back surface lens deposits. |
| | V | isit 1: Treatment 1 Lens Dispensing |
| Step | Procedure | Details |
| 1.26 | Exit VA | Record subjects' distance visual acuity, OD, OS, and OU to the nearest letter. |
| 1.27 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Visual acuity is 20/30 or better OD and OS • The lens fit is acceptable OD and OS • Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 1.28 | Dispense | <ul> <li>The lenses will be dispensed for a 5-9 day wearing period. During this time, they are required to wear the lenses at least 5 days and at least 8 hours per day that they are worn.</li> <li>Dispense enough lenses to last the subject to their scheduled follow-up visit. Do not dispense extras*</li> <li>The lenses will be worn as daily wear/daily disposable only</li> <li>Rewetting drops are permitted if needed</li> <li>A patient instruction booklet will be provided</li> <li>Subjects will be scheduled for their 1-week follow-up visit</li> <li>Subjects should be instructed to wear the study lenses to the follow-up visit and bring their habitual correction with them.</li> </ul> |

| | Visit 1: Treatment 1 Lens Dispensing | |
|---|---|---|
| Step | Procedure | Details |
| | | * Note: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |

VISIT 2
Subjects should attend wearing their study lenses.

| | | sit 2: Treatment 1 Follow-Up Visit |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| 2.2 | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 2.3 | Compliance | Confirm compliance with the prescribed wear schedule. |
| 2.4 | Follow-Up<br>Questionnaires (CLUE) | The subject will respond to the Follow-Up<br>Questionnaire. |
| 2.5 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 2.6 | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 2.7 | Distance ETDRS<br>LogMAR Visual<br>Acuity | Perform monocular distance ETDRS LogMAR visual acuity test at a 4-meter distance over the test eye only under the following conditions: |
| | | <ul> <li>dim illumination (e.g., &lt;2.5 lux), low luminance, with high contrast charts (LLHC)</li> <li>bright illumination (e.g., &gt;400 lux), high luminance with low contrast charts (HLLC)</li> <li>The Precision Vision 4-meter high contrast ETDRS charts (Chart 1 and Chart 2 OD, Chart 3 and Chart 4 OS) and low contrast ETDRS charts (Chart 1 and</li> </ul> |

| | Visit 2: Treatment 1 Follow-Up Visit | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | 2 OD and Chart 3 and Chart 4 OS) will be used. | <del></del> |
| | | Two measurements per condition will be performed. | |
| 2.8 | Subjective Lens Fit | Evaluate overall lens fit acceptance (acceptable or | |
| | Assessment | unacceptable) based on centration, movement and other fitting characteristics. | |
| | | An unacceptable fit is deemed by one of the following criteria: | |
| | | <ul> <li>limbal exposure at primary gaze or with<br/>extreme eye movement</li> <li>edge lift</li> </ul> | |
| | | <ul> <li>excessive movement in primary and up gaze</li> </ul> | |
| | | <ul> <li>insufficient movement in all three of the<br/>following conditions: primary gaze, up<br/>gaze, and Josephson push up</li> </ul> | |
| ė. | | Note: if lens fit is unacceptable subject will be discontinued from the study. | |
| 2.9 | Wettability<br>Characteristics | Record the white light lens wettability of both lenses. | |
| 2.10 | Surface Deposits | Record any front and back surface lens deposits. | |
| 2.11 | Lens Damage | Using the slit lamp, assess lenses for damage. | |
| 2.12 | Lens Removal | The lenses will be removed and stored in the following manner: | |
| | | The OD and OS lenses will be stored wet (using saline solution) in separate glass vials with labels that minimally contain study number, date, subject number, and eye from which the lens was removed in a study specific refrigerator. (Temperature monitoring of refrigerator not required) | |
| | | *The lenses will be shipped back to the Sponsor ambiently once the study has completed. | |
| 2.13 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. | |
| | | Limbal and Bulbar Conjunctival Hyperemia findings and detailed Corneal Staining Assessment will be recorded using a more detailed scale for internal purposes only. Conjunctival hyperemia should be assessed using the 0.5 increment grading scale. | |

| Visit 2: Treatment 1 Follow-Up Visit | | |
|---|---|---|
| Step | Procedure | Details |
| 2.14 | | |
| 2.14 | Eye Rinse | The investigator or technician may rinse the subject's eyes with sterile saline. |
| 2.15 | Visual Acuity | Record the distance Snellen visual acuity with their habitual contact lenses or spectacles (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 2.16 | Instructions | The subject will be instructed to wear their habitual lenses for 7-9 days. |

VISIT 3
Subjects should attend wearing their habitual lenses.

| Visit 3: Post Wash-out Baseline | | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.1 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. | |
| 3.2 | Background PRO<br>Questionnaire (CLUE) | Subject will complete questions regarding their experiences with their habitual lenses. | |
| 3.3 | Contact lens wear times | Record the current wear time (WT) and comfortable wear time (CWT). | |
| 3.4 | Subject-reported Ocular<br>Symptoms | Subject Reported Ocular Symptoms and Problems | in the state of th |
| 3.5 | Distance visual acuity (VA) | Record the distance Snellen VA for OD, OS and OU. Subject must keep reading smaller lines until less than half the letters are correctly identified. | |
| 3.6 | Remove habitual lenses | The subject's habitual lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. | |
| 3.7 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are Grade 3 or higher, the subject is discontinued from the visit as ineligible and may be rescheduled for another baseline visit for the randomization period. | |
| | | Limbal and Bulbar Conjunctival Hyperemia findings and detailed Corneal Staining Assessment will be recorded using a more detailed scale for internal purposes only. Conjunctival hyperemia should be assessed using the 0.5 increment grading | |

| Visit 3: Post Wash-out Baseline | | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | scale. | 50 S |
| 3.8 | Eye Rinse | The investigator or technician may rinse the subject's eyes thoroughly with sterile saline. | |
| 3.9 | Eligibility after Baseline | All responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. One additional baseline examination is permitted to be performed if the subject does not meet the eligibility criteria at the initial baseline visit If subject is deemed to be ineligible after baseline, proceed to Final Evaluation and complete all forms. | |
| 3 | | Visit 3: Treatment 2 Fitting | |
| Step | Procedure | Details | |
| 3.10 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective best sphere refraction. Record the test condition. | |
| 3.11 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. | |
| | | Note: A PIG will be given to the subject in any study where a lens is placed on eye. The subject may wear the study lenses only at the clinical site, or the subjects may be dispensed additional lenses to wear outside of the clinical site. | |
| 3.12 | Lens damage | Using the slit lamp, assess lenses for damage. If any defects are noted, investigator should complete a Product Quality Complaint in EDC. | |
| | | Damaged lenses will be removed and stored in the following manner: The OD and OS lenses will be stored wet (using saline solution) in separate glass vials with labels that minimally contain study number, date, subject number, and eye from which the lens was removed. | |
| | | Replace lens if damaged. | |
| 3.13 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 3.14 | Subjective Best Sphere<br>Over Refraction | Perform subjective best sphere refraction over the study lenses with a phoropter (adopt the maximum | |

| Visit 3: Post Wash-out Baseline | | | |
|---|---|---|--|
| Step | Procedure | Details | |
| | | plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, and OU). | |
| | | Note: The endpoint criterion for the duo-chrome test is the lens power at which the red and green sides of the chart appear to be equally distinct. However, if the subject's response changes from "red" to "green" with only a 0.25D change in power and no report that the two sides appear to be equally sharp, the refraction endpoint should be the lens power that leave the red chart sharper. | |
| 3.15 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is not plano. For each power modification, repeat steps (1.15-1.19). | |
| | | Up to one power modifications are allowed. | |
| 3.16 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 3.17 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. | |
| | | An unacceptable fit is deemed by one of the following criteria: | |
| | | <ul> <li>limbal exposure at primary gaze or with extreme eye movement</li> <li>edge lift</li> <li>excessive movement in primary and up gaze</li> <li>insufficient movement in all three of the</li> </ul> | |
| | | following conditions: primary gaze, up gaze, and Josephson push up Note: if lens fit is unacceptable subject will be | |
| | | discontinued from the study. | |
| 3.18 | Distance ETDRS<br>LogMAR Visual Acuity | Perform monocular distance ETDRS LogMAR visual acuity test at a 4-meter distance over the test eye only under the following conditions: | |
| | | <ul> <li>dim illumination (e.g., &lt;2.5 lux), low luminance, with high contrast charts (LLHC)</li> <li>bright illumination (e.g., &gt;400 lux), high</li> </ul> | |
| Visit 3: Post Wash-out Baseline | | | |
|---|---|---|---|
| Step | tep Procedure Details | | |
| | | luminance with low contrast charts (HLLC) | ia ia |
| | | The Precision Vision 4-meter high contrast ETDRS charts (Chart 1 and Chart 2 OD, Chart 3 and Chart 4 OS) and low contrast ETDRS charts (Chart 1 and 2 OD and Chart 3 and Chart 4 OS) will be used. | |
| | | Two measurements per condition. | |
| 3.19 | White Light Lens<br>Surface Wettability | Record the white light lens wettability of both lenses. | |
| 3.20 | Surface Deposits | Record any front and back surface lens deposits. | |
| | Vis | sit 3: Treatment 2 Lens Dispensing | 7g - 18 |
| Step | Procedure | Details | |
| 3.21 | Exit VA | Record subjects' distance visual acuity, OD, OS, and OU to the nearest letter. | |
| 3.22 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Visual acuity is 20/30 or better OD and OS • The lens fit is acceptable OD and OS • Investigator approval If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. | |
| 3.23 | Dispense | The lenses will be dispensed for a 5-9 day wearing period. During this time, they are required to wear the lenses at least 5 days and at least 8 hours per day that they are worn. • Dispense enough lenses to last the subject to their scheduled follow-up visit. Do not dispense extras* • The lenses will be worn as daily wear/daily disposable only • Rewetting drops are permitted if needed • Subjects will be scheduled for their 1-week follow-up visit and bring their habitual correction with them • Subjects should be instructed to wear the study lenses to the follow-up visit * Note: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to | |

| | Visit 3: Post Wash-out Baseline | |
|---|---|---|
| Step | Procedure | Details |
| | | the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |

VISIT 4
Subjects should attend wearing their study lenses.

| | V | isit 4: Treatment 2 Follow-Up Visit | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.1. | Adverse Events<br>and Concomitant<br>Medications<br>Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | a a |
| 4.2. | Wearing Time | Record the average wearing time and comfortable wearing time. | |
| 4.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 4.4. | Follow-Up<br>Questionnaire<br>(CLUE) | The subject will respond to the Follow-Up<br>Questionnaire. | |
| 4.5. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 4.6. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 4.7. | Distance ETDRS LogMAR Visual Acuity | Perform monocular distance ETDRS LogMAR visual acuity test at a 4-meter distance over the test eye only under the following conditions: • dim illumination (e.g., <2.5 lux), low luminance, with high contrast charts (LLHC) • bright illumination (e.g., >400 lux), high luminance with low contrast charts (HLLC) The Precision Vision 4-meter high contrast ETDRS charts (Chart 1 and Chart 2 OD, Chart 3 and Chart 4 OS) and low contrast ETDRS charts (Chart 1 and 2 OD and Chart 3 and Chart 4 OS) will be used. Two measurements per condition will be performed. | |

| Visit 4: Treatment 2 Follow-Up Visit | | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.8. | Subjective Lens | Evaluate overall lens fit acceptance (acceptable or | |
| 1.0. | Fit Assessment | unacceptable) based on centration, movement and other fitting characteristics. | |
| | | An unacceptable fit is deemed by one of the following criteria: | |
| | | limbal exposure at primary gaze or with<br>extreme eye movement | |
| | | <ul> <li>edge lift</li> <li>excessive movement in primary and up gaze</li> </ul> | |
| | | insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up | |
| | | <u>Note:</u> if lens fit is unacceptable subject will be discontinued from the study. | |
| 4.9. | Wettability<br>Characteristics | Record the white light lens wettability of both lenses. | 100<br>100<br>100 |
| 4.10. | Surface Deposits | Record any front and back surface lens deposits. | |
| 4.11. | Lens Damage | Using the slit lamp, assess lenses for damage. | |
| 4.12. | Lens Removal | The lenses will be removed and stored in the following manner: | |
| | | The OD and OS lenses will be stored wet (using saline solution) in separate glass vials with labels that minimally contain study number, date, subject number, and eye from which the lens was removed in a study specific refrigerator. (Temperature monitoring of refrigerator not required) | |
| | | *The lenses will be shipped back to the Sponsor ambiently once the study has completed. | |
| 4.13. | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. | |
| | | Limbal and Bulbar Conjunctival Hyperemia findings and detailed Corneal Staining Assessment will be recorded using a more detailed scale for internal purposes only. Conjunctival hyperemia should be assessed using the 0.5 increment grading scale. | |
| 4.14. | Eye Rinse | The investigator or technician may rinse the subject's eyes with sterile saline. | |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Step Procedure Details | |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Subjective<br>spherocylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, and OU). |
| F.3 | Comments and<br>Signature | Record any additional information on the page provided and sign the form. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | | |
|---|---|---|---|
| Step | Procedure | dure Details | |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit. | - |
| U.2 | Adverse Events and<br>Concomitant<br>Medications<br>Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. | |
| U.4 | Subjective Sphero-<br>cylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS, and OU). | |
| U.5 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. | |
| U.6 | Dispensing (if applicable) | Subject may be provided with additional lenses as needed to allow continuation in the study if applicable | |
| U.7 | Exit Visual Acuity | Record the subject's exit distance visual acuity (OD, OS, and OU) to the nearest letter. | |

# 7.4. Laboratory Procedures

Not Applicable.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- · provided informed consent
- they are eligible
- · completed all scheduled visits.

# 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

· Subject death during the study period

- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject misses any study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort, or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject.

An additional subject will be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: See Section 3.3

Concomitant therapies that are disallowed include: See Section 3.3

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation

immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site

- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (Refer to for test article return instructions)

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

**Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect, or
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization

- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

# 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events - see definition in Section 13.2.2)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

## 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

# 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)

- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

#### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

# **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.4.3. Event of Special Interest

None

## 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data

will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below. A stand-alone Statistical Analysis Plan (SAP) with more details will be finalized before the interim analysis is undertaken.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

#### 14.2. Sample Size Justification

The plan is to enroll at total of 100 subjects with a target of 90 subjects to complete the study. This is a feasibility study and the sample size was not based on any empirical power calculation. The sample size was considered sufficiently large to gain first insight of the performance of the Test lens with respect to comfort and vision.

There are no historical data available on how the Test lens will perform against the Control lens. Assuming a sample size of 90 subjects, the statistical power was calculated for different scenarios of effect size on CLUE scores ( $\Delta$ ), standard deviation ( $\sigma$ ) and intersubject correlation ( $\rho$ ) using two-sided 5% significance level. The results are summarized below:

Table 5: Statistical Power by effect size, intra-class correlation and standard deviation

| Effect size | Inter-subject | Power (%) $\sigma = 21$ | Power (%) $\sigma = 24$ |
|---|---|---|---|
| $(\Delta)$ | correlation (ρ) | $\sigma = 21$ | $\sigma = 24$ |
| | 0.3 | 50.9 | 37.9 |
| 0 | 0.5 | 65.0 | 49.8 |
| | 0.7 | 85.7 | 71.4 |
| | 0.3 | 84.5 | 69.8 |
| 2.5 | 0.5 | 94.0 | 83.5 |
| | 0.7 | 99.5 | 96.6 |
| | 0.3 | 97.8 | 91.1 |
| 5 | 0.5 | 99.7 | 97.4 |
| | 0.7 | 99.9 | 99.9 |

The power analysis was conducted using the PROC POWER procedure available in SAS for paired tests.

The possible range of standard deviation were considered based on the available historical data summarized below for the Control lens.

Table 6: 1-week CLUE comfort and vision for 1 Day ACUVUE MOIST in historical studies

| | CLUE Comfort | | | CLUE Vision | | |
|-------|--------------|-------|--------|-------------|-------|--------|
| | N | Mean | STD | N | Mean | STD |
| | 66 | 56.38 | 24.655 | 66 | 65.04 | 22.824 |
| | 68 | 63.87 | 24.693 | 68 | 65.17 | 22.110 |
| | 138 | 58.72 | 22.643 | 138 | 61.24 | 20.643 |
| | 142 | 57.21 | 21.341 | 142 | 61.71 | 19.345 |
| | 142 | 60.10 | 26.356 | 142 | 63.52 | 23.652 |
| | 70 | 72.05 | 21.487 | 70 | 72.81 | 20.624 |
| Total | 626 | 60.49 | 23.93 | 626 | 63.99 | 21.67 |

## 14.3. Analysis Populations

## **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Subjects who return to Visits 2 and 4 out of the prescribed visit window will be excluded from the cohort population. Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

### **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

## 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

## 14.5. Primary Analysis

The co-primary endpoints for this study are the CLUE comfort and the CLUE vision scores evaluated after 1-week of lens wear. The primary analysis will be conducted on per-protocol and ITT populations.

### CLUE Comfort and Vision scores

CLUE comfort and vision scores will be analyzed separately using a Bayesian repeated measurement random-effects model to compare between Test and Control lenses. Each regression model will include baseline values, lens type, lens wearing sequence and lens wearing period as fixed effects and investigational site as random effect. Other subject characteristics such as age, gender and will also be included as fixed effects when appropriate. Unstructured covariance matrix will be used to model the residual errors among observations within subjects. Non-informative prior distributions will be used for the coefficients in the models as well as for the error terms. Independent vague normal N(0,1000) priors will be used for the regression coefficients, inverse gamma IG(0.001, 0.001) for the variance of the random effect site and inverse Wishart for the residual errors. The Metropolis sampler algorithm as implemented in the SAS MCMC Procedure will be used to carry out parameter estimation. Results will be reported as regression coefficient mean estimates with credible intervals.

The null and alternative hypotheses for non-inferiority of Test lens relative to Control are as follows:

*H*0:  $\Delta$  < -5 *HA*:  $\Delta$   $\geq$  -5

where  $\Delta$  is the CLUE score mean difference between Test lens and Control lens (Test minus Control). Non-inferiority will be declared if the lower bound of the credible interval of the mean difference between Test and Control is greater than -5.

#### 14.6. Secondary Analysis

# Visual Performance

Monocular distance visual performance in logMAR scale will be analyzed using a Bayesian repeated measurement random-effects model to compare between Test and Control lenses. The regression model will include baseline values, lens type, lens wearing sequence and lens wearing period as fixed effects; and investigational site and patient as random effects. Other subject characteristics such as age, gender and will also be included as fixed effects when appropriate. Unstructured covariance matrix will be used to model the residual errors among observations within same eye and subject across wearing periods. Non-informative prior

distributions will be used for the coefficients in the models as well as for the error terms. Independent vague normal N(0,1000) priors will be used for the regression coefficients, inverse gamma IG(0.001, 0.001) for the variance of the random effect site and inverse Wishart for the residual errors. The Metropolis sampler algorithm as implemented in the SAS MCMC Procedure will be used to carry out parameter estimation. Results will be reported as regression coefficient mean estimates with credible intervals.

The null and alternative hypotheses for non-inferiority of Test lens relative to Control are as follows:

*H*0:  $\Delta > 0.05$  *HA*:  $\Delta \le 0.05$ 

where  $\Delta$  is the mean difference in logMAR between Test lens and Control lens (Test minus Control). Non-inferiority will be declared if the upper bound of the credible interval of the mean difference between Test and Control is less than 0.05.

# Average Daily Wearing Time

Average daily wear time will be analyzed using the same Bayesian model described in the primary analysis.

The null and alternative hypotheses for non-inferiority of Test lens relative to Control are as follows:

*H*0:  $\Delta$  < -1 *HA*:  $\Delta$  > -1

where  $\Delta$  is the mean difference in average daily wearing time between Test lens and Control lens (Test minus Control). Non-inferiority will be declared if the lower bound of the credible interval of the mean difference between Test and Control is greater than -1.

## 14.7. Other Exploratory Analyses

A subgroup analysis will be conducted by considering only subjects who are habitual users of 1 Day ACUVE Moist. Further Bayesian analysis on the primary endpoints will be conducted by incorporating historical control data (see Table 6).

# 14.8. Interim Analysis

No interim analysis is planned.

#### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-

random. To evaluate the impact of missing data, sensitivity analysis may be considered by automatically sampling all missing values and incorporating them in the Markov chain for the parameters using the PROC MCMC procedure.

## 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system from Bioclinica. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Date Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events

- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record. Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source

data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

#### 18. ETHICAL AND REGULATORY ASPECTS

# 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

#### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

### 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject. Each subject for this study will complete an assent and a parent or legal guardian must give written informed consent according to local requirements after the nature of the study has been fully explained. The assent and consent forms must be signed before performance of any study-related activity. The assent and consent forms that are used must be approved by both the Sponsor and by the reviewing IEC/IRB. The assent and informed consent forms should be in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and GCP guidelines, applicable regulatory requirements, and Sponsor policy.

Before entry into the study or pre-screening, the Investigator or an authorized member of the clinical site personnel must explain to the potential subject and parent and/or legal guardian the aims, methods, reasonably anticipated benefits, and potential hazards of the study or pre-screening, and any discomfort it may entail. Subjects and parent and/or legal guardian will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the subject will receive.

Finally, they will be told that the Investigator will maintain a subject identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized Sponsor personnel without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) or regulations. By signing the assent and informed consent form, the subject is authorizing such access and agrees to be

contacted after study completion by health authorities and authorized Sponsor personnel for the purpose of obtaining consent for additional safety evaluations if needed.

## 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or

alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

# 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/4557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html



2

| Protocol 6324 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|

3

6

# APPENDIX B: PATIENT INSTRUCTION GUIDE

To be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

1-DAY ACUVUE® MOIST

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Instruction Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



1-DAY ACUVUE® MOIST Brand Contact Lenses 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses

> etafilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear



**R**Only CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

CR-6324, v 2.0

### SYMBOLS KEY

The following symbols may appear on the label or packaging:

| SYMBOL | DEFINITION |
|-------------------|-----------------------------------------------------|
| (li | Consult Instructions for Use |
| | Manufacturer |
| س | Date of Manufacture |
| $\square$ | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterilized Using Steam Heat |
| 8 | Do Not Re-Use (Single Use) |
| <b>™ ♦</b> | Lens Orientation Correct |
| X X | Lens Orientation Incorrect (Lens Inside Out) |
| <b>C€</b><br>0086 | Quality System Certification Symbol |
| 0 | Fee Paid for Waste Management |
| EC REP | Authorized Representative in the European Community |

Visit www.acuvue.com/guides for additional information about symbols.

### DESCRIPTION

1-DAY ACUVUE® MOIST Brand Contact Lenses, 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM, and 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are soft (hydrophilic) contact lenses available as spherical, toric, or multifocal lenses, and include LACREON® Technology.

The lens material (etaflicon A) is a copolymer of 2-hydroxyethyl methacrylate and methacrylic acid cross-linked with 1, 1, 1-trimethylol propane trimethacrylate and ethylene glycol dimethacrylate.

CR-6324, v 2.0


The lenses are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling. A benzotriazole UV absorbing monomer is used to block UV radiation.

### Lens Properties:

The physical/optical properties of the lens are:

Specific Gravity (calculated): 0.98 – 1.12
 Refractive Index: 1.40
 Light Transmittance: 85% minimum
 Surface Character: Hydrophilic
 Water Content: 58%

Oxygen Permeability (D/k):

VALUE METHOD

21.4 x 10 <sup>11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, edge corrected)

(ml O₂/ml x mm Hg) @ 35°C

28.0 x 10 <sup>11</sup> (cm²/sec) Fatt (boundary corrected, non-edge corrected)

(ml O₂/ml x mm Hg) @ 35°C

Lens Parameters Ranges:

• Diameter (DIA):

Diameter (DIA): 12.0 mm to 15.0 mm
 Center Thickness: Varies with power
 Base Curve (BC): 7.85 mm to 10.00 mm
 Spherical Power (D): -20.00D to +20.00D
 Cylinder Power (CYL): -0.25D to -10.00D
 Axis (AXIS): 2.5° to 180°
 ADD Powers: +0.25D to +4.00D

### **AVAILABLE LENS PARAMETERS**

1-DAY ACUVUE® MOIST Brand Contact Lenses are hemispherical shells of the following dimensions:

Diameter (DIA): 14.2 mm

Center Thickness: 0.084 mm to 0.230 mm (varies with power)

CR-6324, v 2.0 Page 74of 161 JJVC CONFIDENTIAL

Base Curve (BC): 8.5 mm, 9.0 mm

Powers (D): -0.50D to -6.00D (in 0.25D increments)

-6.50D to -12.00D (in 0.50D increments) +0.50D to +6.00D (in 0.25D increments)

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are hemitoric shells of the following dimensions:

Diameter (DIA): 14.5 mm

Center Thickness: 0.090 mm to 0.189 mm (varies with power)

Base Curve (BC): 8.5 mm

Powers (D): +0.00 to -6.00D (in 0.25D increments)

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\* Axis (AXIS): 10° to 180° in 10° increments \*-2.25D cylinder is available in 10°, 20°, 70°, 80°, 90°,

100°, 110°, 160°, 170°, 180° axes only -6.50D to -9.00D (in 0.50D increments)

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\* Axis (AXIS): 10°, 20°, 60°, 70°, 80°, 90°, 100°, 110°,

120°, 160°, 170°, 180°

\*-2.25D cylinder is available in 20°, 90°, 160°, 180°

axes only

+0.25D to +4.00D (In 0.25D increments) Cylinders (CYL): -0.75D, -1.25D, -1.75D

Axis (AXIS): 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are hemispherical shells of the following dimensions:

Diameter (DIA): 14.3 mm

Center Thickness: 0.084 mm to 0.207 mm (varies with power)

Base Curve (BC): 8.4 mm

 Powers (D):
 +6.00D to -9.00D (in 0.25D increments)

 Near ADD Powers (MAX ADD):
 Low Near ADD (LOW): +1.25D Medium Near ADD (MID): +1.75D

High Near ADD (HGH): +2.50D

CR-6324, v 2.0

<sup>4</sup> JJVC CONFIDENTIAL

### TRANSMITTANCE CURVES

1-DAY ACUVUE® MOIST Brand Contact Lenses (etaflicon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



 $^{\circ}$ The data are representative measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-3.00D lens, 0.084 mm center thickness).

 Lerman, S., Radiant Energy and the Eye, MacMilan, New York, 1980, p. 58, figure 2-21
 Waxler, M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

### **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays on the retina.

The UV Blocking for these lenses averages 97% in the UVB range of 280 nm to 315 nm and 82% in the UVA range of 316 nm to 380 nm for the entire power range.

CR-6324, v2.0


NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

### INDICATIONS (USES)

- 1-DAY ACUVUE® MOIST Brand Contact Lenses are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1.00D or less of astigmatism.
- 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 0.50D to 3.00D of astigmatism.
- 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are indicated for daily disposable wear for the optical correction of distance and near vision in presbyopic phakic or aphakic persons with non-diseased eyes who may have 4,00D of ADD power or less and 0,75D or less of astigmatism.

The lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

When prescribed for daily disposable use, no cleaning or disinfection is required. Lenses should be discarded upon removal.

### CONTRAINDICATIONS (REASONS NOT TO USE)

DO NOT USE these lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye.
- Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.
- · Severe insufficiency of lacrimal secretion (dry eye).
- Corneal hypoesthesia (reduced corneal sensitivity).

CR-6324,v2.0

<sup>6</sup> JJVC CONFIDENTIAL

- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocular irritation due to allergic reactions which may be caused by use
  of contact lens solutions (i.e., rewetting drops) that contain chemicals or
  preservatives (such as mercury, Thimerosal, etc.) to which some people
  may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral).
- If eyes become red or irritated.

### WARNINGS

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION. IF THE PATIENT EXPERIENCES:

- · Eye Discomfort,
- · Excessive Tearing,
- · Vision Changes,
- . Loss of Vision,
- · Eye Redness, or
- Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

- When prescribed for daily wear, patients should be instructed not to wear their lenses while sleeping. Clinical studies have shown that when lenses are worn overnight, the risk of ulcerative keratitis is greater than among those who do not wear them overnight.<sup>3</sup>
- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.

CR-6324, v2.0


 The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

<sup>3</sup> New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

### Specific Instructions for Use and Warnings:

Water Activity

Instruction for Use

Do not expose contact lenses to water while wearing them.

### WARNING

Water can harbor microorganisms that can lead to severe infection, vision loss, or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

### **PRECAUTIONS**

### Special Precautions for Eye Care Professionals:

 Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.

 Patients who wear these lenses to correct presbyopia using monovision (or modified monovision using 1-DAY ACUVUE® MOIST Brand MULTIFOCAL) may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.

CR-6324, v 2.0


- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove lenses immediately if the eyes become red or irritated.

# Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

### **Handling Precautions:**

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- . DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup.
- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the Patient Instruction Guide for these lenses and those prescribed by the Eye Care Professional.
- · Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container. Slide the lens up the side of the bowl until it is free of the container.
- Do not touch the lens with fingernalls.

### Lens Wearing Precautions:

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for Sticking (Non-Moving) Lenses." The lens should move freely on the eye for the continued health of the eye. If nonmovement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.

9

- . The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- · If aerosol products, such as hairspray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and furnes while wearing lenses.

### Lens Care Precautions:

. The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

### Other Topics to Discuss with Patients:

- · Always contact the Eye Care Professional before using any medicine in the eyes.
- · Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- · As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

### Who Should Know That the Patient is Wearing Contact Lenses?

- · Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- · Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

### **ADVERSE REACTIONS**

The patient should be informed that the following problems may occur when wearing contact lenses:

- · The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, comeal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.

CR-6324, v 2.0

Page 82 of  $161^{11}$ JJVC CONFIDENTIAL

### **GENERAL FITTING GUIDELINES**

### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- Motivation to wear lenses
- Ability to follow instructions regarding lens wear
- General health
- · Ability to adequately handle and care for the lenses
- · Ability to understand the risks and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses

### B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the lens fitting instructions as outlined below.

### C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4.00D.

### D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, corneal curvature measurements should be performed to establish the patient's baseline ocular status.

CR-6324, v2.0 p.


- 1-DAY ACUVUE® MOIST: 8.5 mm/14.2 mm
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: 8.5 mm/14.5 mm
- 1-DAY ACUVUE® MOIST MULTIFOCAL: 8.4 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

### 1. Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

### 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

### 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

### E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

1.

CR-6324, v2.0 


| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |
| Example 2 | |
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |
| Final lens power: | -1.75D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see **PATIENT MANAGEMENT** section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### **TORIC FITTING GUIDELINES**

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing 1-DAY ACUVUE® MOIST for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the patient.

### A. How to Determine Lens Cylinder and Axis Orientation

### 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position – there is no "top" and "bottom" as in a prism-ballasted lens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.

14

CR-6324, v2.0




You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

### 3. Assessing Rotation

imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift," measure or estimate the "drift," then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.

15

CR-6324, v 2.0


### B. Final Lens Power

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

### 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx > 4.00D, compensate for vertex distance. If sphere alone or combined sphere and cylinder  $Rx \le \pm 4.00D$ , vertex compensation is not necessary.

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq$  0.50D from the refractive cylinder.

### 3. Case Examples

### Example 1

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20 O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis 180°. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx prescribed:

O.D. -2.50D / -1.25D x 180°

O.S. -2.00D / -0.75D x 180°

 JJVC CONFIDENTIAL CR-6324, v 2.0

### Example 2

Manifest (spectacle) refraction: O.D. -3.00D / -1.00D x 90° 20/20 O.S. -4.75D / -2.00D x 90° 20/20

Choose diagnostic lenses of  $-3.00D/-0.75D \times 90^\circ$  for the right eye and  $-4.50D/-1.75D \times 90^\circ$  for the left eye, the nearest lenses available to the spherical power and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

### Right Eye

The orientation mark on the right lens rotates left from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx prescribed: O.D. -3.00D / -0.75D x 100°

### Left Eve

The orientation mark on the left lens rotates right from the 6 o'clock position by  $10^\circ$  and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate for the 10° axis drift by subtracting it from the manifest refraction axis.

Here is the Rx prescribed: O.S. -4.50D / -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see **PATIENT MANAGEMENT** section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

CR-6324, v 2.0 Page 88 of <sup>17</sup>161 JJVC CONFIDENTIAL

### **MULTIFOCAL FITTING GUIDELINES**

### A. Presbyopic Needs Assessment & Patient Education

Multifocal contact lenses may produce compromise to vision under certain circumstances and the patient should understand that they might not find their vision acceptable in specific situations (i.e., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments. Occupational and environmental visual demands should be considered. If the patient requires critical visual acuity and stereopsis, it should be determined by trial whether this patient can function adequately with 1-DAY ACUVUE\* MOIST MULTIFOCAL. Wearing these lenses may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet their state driver's license requirements with the 1-DAY ACUVUE® MOIST MULTIFOCAL should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

1-DAY ACUVUE® MOIST MULTIFOCAL is not recommended for patients who have -1.00D or greater of refractive cylinder as this level of uncorrected cylinder may lead to additional visual compromise. These lenses are available in the following ADD powers:

- Lens "LOW" = low near ADD lens (Max ADD +1.25)
- Lens "MID" = medium near ADD lens (Max ADD +1.75)
- Lens "HGH" = high near ADD lens (Max ADD +2.50)

### B. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4.00D. Determine the spherical equivalent distance prescription for a muttifocal patient. Determine the eye dominance using one of the methods below:

18 JJVC CONFIDENTIAL

 $CR\text{-}6324,\,v\;2.0\qquad \text{}$ 

Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2 Determine which eye does not accept added plus power. Place a +1.00D hand-held trial lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes while the patient is viewing the distance visual acuity chart. The eye with the plus over it that the patient notices the greatest reduction in vision is determined to be the dominant eye.

### C. Select the Initial Trial Lens

- For each eye, select the trial lens distance power that is closest to the
  patient's distance spherical equivalent. Remember to compensate for
  vertex distance if the refraction is greater than ±4.00D.
- Select the near power of the lens based on the patients ADD range as follows:
  - ADD: +0.75D to +1.25D use a low near ADD (LOW) lens on each eye
  - ADD: +1.50D to +1.75D use a medium near ADD (MID) lens on each eye
  - ADD: +2.00D to +2.50D use a medium near ADD (MID) on the dominant eye and a high near ADD (HGH) lens on the non-dominant eye
- 3. Allow the lenses to settle for a minimum of 10 minutes.
- 4. Assess distance and near vision binocularly and monocularly.
- Demonstrate the vision under various lighting conditions (normal and decreased illumination) and at distance, intermediate, and near.
- Make adjustments in power as necessary based on the distance overrefraction. The use of hand-held trial lenses is recommended. Check the impact on distance and near vision.
- 7. If vision is still unacceptable, make adjustments in power as necessary (see "Multifocal Troubleshooting" below). If distance and near vision are acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).


### D. Multifocal Troubleshooting

### Unacceptable Near Vision

If it has been determined that no change is required based on the overrefraction, then add +0.25D to the spherical power of the non-dominant eye.

### Unacceptable Distance Vision

If it has been determined that no change is required based on the overrefraction, then make the changes as listed below:

- If the patient is wearing two "LOW" ADD lenses, change the dominant eye to a 1-DAY ACUVUE® MOIST sphere lens with a power equal to the spherical equivalent distance prescription.
- If the patient is wearing two "MID" ADD lenses, change the ADD power in the dominant eye to the "LOW" ADD power.
- If the patient is wearing a "MID" ADD lens in the dominant eye and a "HGH" ADD lens in the non-dominant eye, change the non-dominant eye to a "MID" ADD lens and add +0.25D to the distance power.

### E. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

CR-6324, v 2.0


### MONOVISION FITTING GUIDELINES

### A. Patient Selection

### 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet their state driver's license requirements with monovision correction should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dimly lit restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision, and straight ahead and upward gaze that monovision contact lenses provide.

### B. Eye Selection

### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2 Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

### 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

### Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

### Visual Demands Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

### C. Special Fitting Characteristics

### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral myope would require corrective lenses on both eyes.

CR-6324, v 2.0


### Examples:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left eye uncorrected for near.

### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the **GENERAL**FITTING GUIDELINES for base curve selection described in this Package Insert.

Case history and a standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next, determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernalis. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

### D. Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact tenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- · Make use of proper illumination when carrying out visual tasks.

Monovision fitting success can be improved by the following suggestions:

- · Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- · Emphasize the benefits of clear near vision, and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### PATIENT MANAGEMENT

- . Follow the accepted standard of care in fitting and following up with your patient, e.g., American Optometric Association standard of care.
- · Schedule the appropriate follow-up examination.
- · Preferably, at the follow-up visits, lenses should have been worn for at least six hours.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses, which can be found at www.acuvue.com. REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

### WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to over wear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

CR-6324, v 2.0


The maximum suggested wearing time for these lenses is:

| DAY | HOURS |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

### REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removel

When disposed of after a single daily use, these lenses may reduce the risk of developing giant papillary conjunctivitis.<sup>4</sup>

When worn as a daily disposable lens, these lenses may provide improved comfort for many patients who experience mild discomfort and itching associated with allergies during contact lens wear, compared to lenses replaced at intervals of greater than 2 weeks.

Clinical research has shown that when worn on a daily disposable basis, these lenses may provide improved comfort for 2 out of 3 patients who reported suffering from discomfort associated with allergies during contact lens wear.

<sup>4</sup>The CLAO Journal, July 1999, Volume 25, Number 3

### LENS CARE DIRECTIONS

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have replacement lenses or spectacles available.

For complete information concerning contact lens handling and care, refer to the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### Care for Sticking (Non-Moving) Lenses

During removal, if the lens sticks to the eye, the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution

26


directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should **immediately** consult the Eye Care Professional.

### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

### **HOW SUPPLIED**

Each UV-absorbing sterile lens is supplied in a foll-sealed plastic package containing buffered saline solution with povidone. The plastic package is marked with the following:

- 1-DAY ACUVUE® MOIST: base curve, power, diameter, lot number, and expiration date
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: base curve, power, diameter, cylinder, axis, lot number, and expiration date
- 1-DAY ACUVUE® MOIST MULTIFOCAL: base curve, power, diameter, ADD power, lot number, and expiration date

### REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with these lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acutus.com

27


Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com



©Johnson & Johnson Vision Care, Inc. 2017 In Canada: Johnson & Johnson Vision Care division of Johnson & Johnson Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed in USA Revision date: 07/17 Revision number: M-07-17-02

> 1-DAY ACUVUE® MOIST and LACREON® are Trademarks of Johnson & Johnson Vision Care, Inc.


# APPENDIX D: LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING LENS FITTING CHARACTERISTICS SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS BIOMICROSCOPY SCALE DISTANCE AND NEAR VISUAL ACUITY EVALUATION DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE PATIENT REPORTED OUTCOMES WHITE LIGHT LENS SURFACE WETTABILITY VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

## LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS

# Limbal & Conjunctival (Bulbar) Redness












# EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING

# **Expanded Sodium Fluorescein Corneal Staining**







# LENS FITTING CHARACTERISTICS













# SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS

# **Subject Reported Ocular Symptoms/Problems**

# FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE











# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS





























# DISTANCE AND NEAR VISUAL ACUITY EVALUATION








## DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE







### PATIENT REPORTED OUTCOMES



#### WHITE LIGHT LENS SURFACE WETTABILITY



# VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING











#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6324 Clinical Evaluation of etafilcon A Contact Lenses

Using a Novel Manufacturing Technology

Version and Date: v2.0, Amendment 1.0 April 26, 2019

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal<br>Investigator: | | |
|----------------------------|------------------------------------------|------|
| _ | Signature | Date |
| | Name and Professional Position (Printed) | • |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | - |